CLINICAL TRIAL: NCT05590741
Title: An Idiographic Examination of Treatment Mechanisms in Emotion Regulation Therapy: A Multiple Case-Based Design
Brief Title: An Idiographic Examination of Treatment Mechanisms in Emotion Regulation Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Principal Investigator, Douglas Mennin, Professor of Clinical Psychology, Director of Clinical Training, Teachers College, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-008
Record Dates: First submitted 2022-10-13; First posted 2022-10-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Rumination; Worry; Self-Criticism; Anxiety; Depression; Distress, Emotional
Keywords: Worry; Rumination; Self-Criticism; Emotion Regulation Therapy; Emotion Regulation; Treatment Mechanisms
MeSH Terms: conditions — Rumination Syndrome; Anxiety Disorders; Depression; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All participants will receive a 12-session version of Emotion Regulation Therapy delivered weekly via synchronous telehealth using videoconferencing software and an asynchronous Internet-based online platform to supplement the content covered in each session.
  Interventions: Behavioral: Emotion Regulation Therapy via Telehealth

INTERVENTIONS:
Behavioral: Emotion Regulation Therapy via Telehealth — The initial stage of treatment focuses on psychoeducation about anxiety/depression, the impact that these cognitions/behaviors/emotions have on recent situations, and self-monitoring of worry/anxiety/depression. The sessions focus on the development of skills that help understand and regulate one's emotional experience (i.e., recognizing emotions when they are happening, identifying the meaning of a given emotion experience, soothing oneself in the context of negative emotional experiences). Following the development of these skills, sessions focus on the application of somatic awareness and emotion regulation skills while imagining emotionally evocative themes. The remaining session focuses on terminating therapy, relapse prevention, and future goals. An Internet-based online platform will be used to promote engagement with and increase accessibility to between-session skills practice and treatment-related activities (e.g., self-monitoring, session summaries, worksheets).
  Other Names: Emotion Regulation Therapy (ERT)

SUMMARY:
This study is an open trial designed to examine individual changes that occur before, during, and after 12 sessions of Emotion Regulation Therapy (ERT) delivered via telehealth for individuals in New York State who are experiencing elevated worry, rumination, or self-criticism.

DETAILED DESCRIPTION:
The main questions this study aims to answer are to:

1. Examine temporal patterns of ERT-specific treatment mechanisms (attention regulation, metacognitive regulation, motivation regulation, and valued living), relationships between these mechanisms and negative self-referential processing (NSRP; i.e., rumination, worry, and self-criticism) severity over time, and changes in these mechanisms in response to specific intervention strategies/modules.
2. Investigate the effect of concordance and/or discordance between therapists and clients regarding skill acquisition, treatment goals, and case conceptualizations on treatment mechanisms as well as measures of treatment outcome and satisfaction.
3. Demonstrate the preliminary efficacy of a 12-session version of ERT in reducing symptoms of psychological distress (e.g., anxiety, depression, worry, rumination, self-criticism), changing ERT-specific treatment mechanisms (e.g., attention regulation), and improving quality of life and overall functioning.

Participants will:

1. Fill out an online pre-screening questionnaire and complete a structured clinical interview via Zoom Healthcare
2. Be enrolled as a patient at the Dean Hope Center for Educational and Psychological Services (DHCEPS), located at Teachers College
3. Attend 12 once-weekly telehealth ERT sessions
4. Complete 18 weekly questionnaires online via Qualtrics (two before starting treatment, 12 each week during treatment, and 4 after ending treatment).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65
* Fluent in English (and therefore able to provide consent)
* Currently living in New York State
* Access to at least one device with internet and video-conferencing capabilities
* High self-reported worry, rumination, and/or self-criticism
* Meet Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for at least one, current psychological disorder

Exclusion Criteria:

* Active suicidal ideation or intent
* Substance dependence disorder, schizophrenia, bipolar-I disorder, or a primary DSM-5 diagnosis of borderline or narcissistic personality disorder
* Currently in therapy or receiving any type of psychosocial treatment
* Individuals taking psychotropic mediation that has not been stabilized for a period of at least 3 months
* Current students at Teachers College, Columbia University

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Weekly Assessment of Change in Attentional Control | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Attentional Control Scale (ACS) is a 21-item measure used to measure difficulties with concentration associated with problems regulating emotions. The focusing and shifting subscales of the ACS align with the two attention emotion regulation (ER) skills taught in ERT.
Weekly Assessment of Change in Decentering | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The decentering subscale of the Experiences Questionnaire (EQ-D) is an 11-item subscale assessing one's ability to distance themselves from their emotional experience, which is one metacognitive ER skill taught during ERT. Higher scores on this subscale indicate better ability to distancing oneself from one's emotional experience.
Weekly Assessment of Change in Reappraisal | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The reappraisal subscale of the Emotion Regulation Questionnaire (ERQ) is a 6-item measure of the ability to regulate emotions, using the strategy of reappraisal. Higher scores on this subscale indicate a better ability to regulate emotions using the strategy of reappraisal.
Weekly Assessment of Change in Valued Living/Action | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Valuing Questionnaire (VQ) is a 10-item measure of the degree to which patients live by their values in daily life. It uses a 7-point Likert scale (0-6) to assess progress and obstructions to valued living. Higher scores on this measure indicate more valued living.
Weekly Assessment of Change in Clarity of Approach-Avoidance Motivation | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Mental Representation of Approach Avoidance Questionnaire (MRAAQ) is a 42-item self-report assessment designed to capture the mental representation of approach-avoidance motivation.

SECONDARY OUTCOMES:
Weekly Assessment of Change in Depression Severity | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v. 1.0 - Emotional Distress - Depression - Short Form 8a will be administered to assess for depression severity. Higher scores on this measure indicate greater depression severity.
Weekly Assessment of Change in Anxiety Severity | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank - Emotional Distress - Anxiety - Short Form 8a will be administered to assess for anxiety severity. Higher scores on this measure indicate greater anxiety severity.
Weekly Assessment of Change in Rumination | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Rumination-Reflection Questionnaire (RRQ) is a 12-item measure that assesses past-focused rumination with specificity regarding the types of rumination that people may experience. Higher scores on this measure indicate greater rumination.
Weekly Assessment of Change in Worry | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Penn State Worry Questionnaire - Past Week (PSWQ-PW) is an adapted version of the original PSWQ, contains 15 items (rated on a 0-6 scale), and assesses the extent to which worry has been excessive, uncontrollable, and pervasive in the past week. Higher scores on this measure indicate greater worry in the past week.
Weekly Assessment of Change in Self-Criticism | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The self-judgment subscale of the Self-Compassion Scale (SCS) contains 5-items and assesses the tendency to self-criticize. Higher scores on this measure indicate greater self-criticism.

OTHER OUTCOMES:
Weekly Assessment of Change in Disability/Impairment | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Sheehan Disability Scale (SDS) is a 4-item scale which assesses impairment in work, social life/leisure activity, family life/home responsibilities, and overall functioning. Higher scores on this measure indicate greater impairment.
Weekly Assessment of Change in Life Satisfaction | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Brief Multidimensional Students' Life Satisfaction Scale (BMSLSS) is a 5-item scale assessing a participant's satisfaction within a number of domains regarding their social and occupational functioning. Higher scores on this measure indicate greater life satisfaction.
Weekly Assessment of Change in Behavioral Regulation | Weekly from Baseline (2 weeks) through Treatment (12 weeks) and Follow-Up (4 weeks)
  The Behavior Regulation Scale (BRS) is a 24-item self-report measure of behaviors engaged for the purposes of ER.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Mennin, Principal Investigator — Professor of Clinical Psychology
Locations (1):
- Teachers College, Columbia University, New York, New York, United States